CLINICAL TRIAL: NCT04890041
Title: Efficacy of TPO-RA in the Management of Primary Immune Thrombocytopenia (ITP) in Patients Older Than 14 Years With Poor First-line Response: a Multi-center, Prospective, One-arm Study
Brief Title: TPO-RA in Primary Immune Thrombocytopenia (ITP) in Patients Older Than 14 Years
Acronym: ITP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020033
Record Dates: First submitted 2021-05-12; First posted 2021-05-18 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2024-10

CONDITIONS: Primary Immune Thrombocytopenic Purpura

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): 100 subjects will be enrolled with the indicated treatment dose of TPO-RA
  Interventions: Drug: TPO-RA

INTERVENTIONS:
Drug: TPO-RA — The subjects will receive an initial dose of TPO-RA once daily. Platelet counts were collected weekly until week 6 of the study. Dosage was adjusted to maintain platelet levels between 50×10^9/L and 150×10^9/L according to platelet count. TPO-RA was administered once a day for 4 weeks. If the platelet count dose not reach 30×10^9/L, the treatment was stopped. If the platelet count is more than 400×10^9/L after taking TPO-RA once a day for 2 consecutive weeks, the treatment will be stopped.
  Other Names: TPO-RAs

SUMMARY:
This multi-center study aims to study the efficacy of TPO-RAs' transformation in Chinese ITP patients older than 14 years. This study will be conducted in ITP patients who had not responded to first-line in the previous treatment .

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the efficacy of TPO-RAs' transformation in Chinese ITP patients older than 14 years who had not responded to first-line in the previous treatment.

100 eligible subjects will be enroll ed in this study.The dose will be adjusted according to the subject platelet count during the period from week 1 to week 6.

ELIGIBILITY:
Inclusion Criteria:

* Men and women greater than or equal to 14 years of age.
* Participants diagnosed with primary immune thrombocytopenia with two platelet counts of < 30x10^9/L or with bleeding at least 7 days apart，do not have evidence of other causes of thrombocytopenia (e.g.,pseudothrombocytopenia, myeloid fibrosis).
* Previous treatment with poor response to first-line therapy and any of the maximum 4-week doses of eltrombopag, herombopag, avatrombopag, or 300U/kg/ day × 14-day rhTPO with no response to treatment (platelet count < 30×109/L after treatment, or platelet count increase less than twice the baseline value, or with bleeding)
* Participants willing and able to comply with the requirements of the study protocol, and sign the informed consent.

Exclusion Criteria:

* Patients diagnosed with secondary immune thrombocytopenia.
* A history of arteriovenous thrombosis, disseminated intravascular coagulation, myocardial infarction, cerebral obstruction, thrombotic microangiopaemia, autoimmune diseases, malignant tumors, liver cirrhosis and other diseases that were not eligible for inclusion.
* Liver disease with one of the following indicators: a. total bilirubin ≥ 2 times of the upper limit of normal; b. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≥ 2 times the upper limit of normal value; Patients with renal disease (serum creatinine ≥ 1.5 times the upper limit of normal);
* Subjects with known allergies to eltrombopag, herombopag, rh-TPO, avatrombopag, or any of excipients;
* Have used rituximab in the past 3 months;
* Splenectomy in recent 3 months;
* Those who are not considered suitable for this study by the researcher;
* Women who are pregnant or who intend to become pregnant in the near future are excluded.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-30 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment response | From the start of study treatment (Day 1) up to the end of week 6
  Percentage of participants whose platelet count achieving response (R) within 6weeks.

SECONDARY OUTCOMES:
Treatment response | From the start of study treatment (Day 1) up to the end of week 1,2, 3, 4, 5 and 6.
  Percentage of participants achieving a platelet count >=50×10^9/L at week 1,2,3,4,5and 6 of treatment.
Treatment response | From the start of study treatment (Day 1) up to the end of week 1,2, 3, 4, 5 and 6.
  Percentage of participants achieving a platelet count >=100×10^9/L at week 1,2,3,4,5and 6 of treatment.
Duration of response | From the start of study treatment (Day 1) up to the end of week 6
  Percentage of participants whose platelet count achieving persistence response (R) within 6weeks(defined as the proportion of subjects with a platelet count of ≥30×109/L for at least 4 weeks of the 6-week treatment period without remedial therapy).
Concomitant medication | From the start of study treatment (Day 1) up to the end of week 6
  The percentage of patients with reduced concomitant medication, reduced bleeding and remedial treatment.
Adverse events | From the start of study treatment (Day 1) up to the end of week 6
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No